CLINICAL TRIAL: NCT00631943
Title: An Open Label, Non-comparative, Multicentre Study to Evaluate the Efficacy and Tolerability of Pregabalin in Peripheral Neuropathic Pain
Brief Title: A Study to Evaluate the Efficacy and Safety of Pregabalin (Lyrica) for the Treatment of Nerve Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081068
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-04

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pregabalin (Lyrica)

INTERVENTIONS:
Drug: Pregabalin (Lyrica) — Oral pregabalin (Lyrica) capsules, initial dose of 75 mg twice daily, which could be increased to 300 mg twice daily at the discretion of the investigator. Patients were treated for up to 21 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Lyrica in Indian patients with nerve pain

ELIGIBILITY:
Inclusion criteria:

* Peripheral neuropathic pain
* Score of at least 40 mm on the VAS of the SF-MPQ at screening and baseline
* Completion of at least 4 daily pain diary entries with an average daily pain score of at least 4 over the 7 days prior to baseline

Exclusion criteria:

(none)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-11; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Short Form McGill Pain Questionnaire (SF-MPQ) visual analog score (VAS) | Weeks 1 and 2 and end of treatment
Change from baseline in weekly mean pain scores | Weeks 1 and 2 and end of treatment

SECONDARY OUTCOMES:
Change from baseline in Euro Quality of Life Questionnaire (EQ-5D) scores | End of treatment
Adverse events and laboratory value changes | Weeks 1 and 2 and end of treatment
Change from baseline in weekly mean sleep interference score | Weeks 1 and 2 and end of treatment
Change from baseline in sensory, affective, and total components of the pain descriptor score and the Present Pain Intensity (PPI) of the SF-MPQ | Weeks 1 and 2 and end of treatment
Change from baseline in Patient Global Impression of Change (PGIC) | Weeks 1 and 2 and end of treatment
Change from baseline in Clinical Global Impression of Change (CGIC) | Weeks 1 and 2 and end of treatment
Change from baseline in pain interference scores on the Brief Pain Inventory (BPI ) Short-Form | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Bangalore, Karnataka / India
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Maharashtra, Mumbai
  - Pfizer Investigational Site, Chennai, Tamil Nadu

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081068&StudyName=A%20study%20to%20evaluate%20the%20efficacy%20and%20safety%20of%20Lyrica%20for%20the%20treatment%20of%20nerve%20pain